CLINICAL TRIAL: NCT04197583
Title: Boston Scientific Double-J PLUS Ureteral Stent Postmarket Patient Registry
Brief Title: Double-J PLUS Postmarket Registry
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: U0652
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Ureter Obstruction
MeSH Terms: conditions — Ureteral Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Boston Scientific Ureteral Stents, Urinary Diversion Stent — A BSC Ureteral Stent is an implantable device that is used to restore flow of urine from the kidney to the bladder in obstructed ureters. A BSC Urinary Diversion Stent is an implantable device that is used to restore flow of urine from the kidney.

SUMMARY:
A multi-center global registry to obtain post-market safety and efficacy data on Boston Scientific Ureteral and Urinary Diversion Stents

ELIGIBILITY:
Inclusion Criteria (for all Ureteral stent types except Urinary Diversion Stents):

* Subject is undergoing placement of a Boston Scientific Ureteral Stent
* Subject anatomy is appropriate to accommodate a stent size available in the study
* Subject is able to accurately detect and report bladder function and pain
* Subject is willing and able to:

  * Complete patient QoL questionnaire at specified time points (for subjects aged ≥ 18 years)
  * Return for all follow-up visits

Inclusion Criteria (for Urinary Diversion Stents):

* Subject is undergoing placement of a Boston Scientific Urinary Diversion Stent(s)
* The anatomical features of the involved renal collecting system are known by either prior or concurrent urography or axial CT imaging
* Subject is willing and able to return for all follow-up visits

Exclusion Criteria (for Ureteral stents and Urinary Diversion Stents):

* Subjects who meet any of the contraindications per individual stent DFU
* Subjects receiving different stent type in case of bilateral/multiple stenting
* Subjects with an indwelling ureteral stent(s) not planned to be removed prior to/or concurrently with the study stent implant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study will enroll patients who are receiving a Boston Scientific Ureteral stent or Urinary Diversion Stent as part of their standard of care.
Sampling Method: Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Krambeck, Principal Investigator — Northwestern University; Michael Borofsky, Principal Investigator — University of Minnesota
Locations (10):
- United States (7):
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - Northwestern University-Department of Urology, Chicago, Illinois
  - NorthShore University HealthSystem, Glenview, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - New York Presbyterian Hospital-Columbia University Medical Center, New York, New York
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
- Vancouver General Hospital, Vancouver, British Columbia, Canada
- Centre Hospit Prive St Gregoire Vivalto, Saint-Grégoire, France
- Nagoya City University Hospital, Nagoya, Aichi-ken, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were generally recruited from physician's practice and met the indications for a ureteral stent implant per the IFU/DFU. Any subject who intended to receive BSC Ureteral Stent(s) as part of their standard of care and was willing to provide a written informed consent was approached and considered for enrollment in the study.
Pre-assignment Details: This section is not applicable.
Groups:
- Boston Scientific Tria Ureteral Stents: Subjects were treated with Tria Boston Scientific Ureteral Stent(s). Subjects were generally recruited from physician's practice and met the indications for a ureteral stent implant per the IFU/DFU. Any subject who intended to receive BSC Ureteral Stent(s) as part of their standard of care and was willing to provide a written informed consent was approached and considered for enrollment in the study.
- Boston Scientific Non- Tria Ureteral Stents: Subjects were treated with Non-Tria Boston Scientific Ureteral Stent(s). Subjects were generally recruited from physician's practice and met the indications for a ureteral stent implant per the IFU/DFU. Any subject who intended to receive BSC Ureteral Stent(s) as part of their standard of care and was willing to provide a written informed consent was approached and considered for enrollment in the study.
Period: Overall Study
Arm/Group | Boston Scientific Tria Ureteral Stents | Boston Scientific Non- Tria Ureteral Stents
Started | 215 | 164
Completed | 162 | 131
Not Completed | 53 | 33
Not completed — Study Stent Replacement | 34 | 8
Not completed — Lost to Follow-up | 14 | 3
Not completed — Death | 3 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Discontinued. Patient had disseminated metastatic condition | 0 | 1
Not completed — Screen Failure | 0 | 20

BASELINE CHARACTERISTICS:
Population: 20 Non-Tria subjects were screen failures and did not complete the Index Procedure.
Groups:
- Boston Scientific Ureteral Stents - Tria: Subjects were treated with Tria Boston Scientific Ureteral Stent(s). Subjects were generally recruited from physician's practice and met the indications for a ureteral stent implant per the IFU/DFU. Any subject who intended to receive BSC Ureteral Stent(s) as part of their standard of care and was willing to provide a written informed consent was approached and considered for enrollment in the study.
- Boston Scientific Ureteral Stents - Non-Tria: Subjects were treated with non-Tria Boston Scientific Ureteral Stent(s). Subjects were generally recruited from physician's practice and met the indications for a ureteral stent implant per the IFU/DFU. Any subject who intended to receive BSC Ureteral Stent(s) as part of their standard of care and was willing to provide a written informed consent was approached and considered for enrollment in the study.
- Total: Total of all reporting groups
Arm/Group | Boston Scientific Ureteral Stents - Tria | Boston Scientific Ureteral Stents - Non-Tria | Total
Number analyzed (Participants) | 215 | 144 | 359
Age, Continuous [Mean (Full Range); unit: years] | 57.2 [19 to 90] | 60.0 [23 to 85] | 58.4 [19 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 58 | 157
  Male | 116 | 86 | 202
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 29 | 18 | 47
  United States | 166 | 98 | 264
  Japan | 20 | 0 | 20
  France | 0 | 28 | 28
Quality of Life Endpoint - Patient-Reported Outcomes [Mean (Full Range); unit: units on a scale] — Pain Interference 6b: score range is 41.0 to 78.3; with higher values being worse quality of life.
  Pain Intensity 3a: score range is 30.7 to 71.8; with higher values being worse quality of life.
  units on a scale
    Patient Reported Outcomes Measurement Information System (PROMIS) Pain Intensity 3a | 44.34 [30.7 to 71.8] | 43.15 [30.7 to 71.8] | 43.86 [30.7 to 71.8]
    Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference 6b | 55.09 [41.0 to 78.2] | 53.85 [41.0 to 78.2] | 54.59 [41.0 to 78.2]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Implanted Stents Meeting the Technical Success Criteria
Description: Technical success was defined as: a stented kidney drains (to bladder) during the planned indwell time with no re-intervention due to obstruction of the stented ureters.
Time Frame: 2 months to 15 Months
Population: Subjects who provided consent and for whom a Boston Scientific stent placement procedure was initiated were included. Number of units analyzed are stents implanted for more than 12 hours. Results were summarized by Tria and Non-Tria separately. Performance goal was 85% for Tria stone management.
Measure: Count of Units; unit: Stent Implanted
Units Other Than Participants: Stent Implanted
Arm/Group | Boston Scientific Ureteral Stents - Tria | Boston Scientific Ureteral Stents - Non-Tria
Number analyzed (Participants) | 215 | 144
Number analyzed (Stent Implanted) | 246 | 160
Stent Implanted
  Technical Success Criteria Met | 242 | 158
  Technical Success Criteria Not Met | 4 | 2
Statistical Analysis 1: Comparison: Boston Scientific Ureteral Stents - Tria vs Boston Scientific Ureteral Stents - Non-Tria; Test type: Other; Proportion by group = 0.984, 95% CI 2-sided [0.948 to 0.995] — For Tria subjects with stone management indication only

2. Primary Outcome: Primary Safety Endpoint
Description: Any Serious Adverse Device Effects
Time Frame: 2 months to 15 Months
Population: Subjects who provided consent and for whom a Boston Scientific stent placement procedure was initiated were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Boston Scientific Ureteral Stents - Tria | Boston Scientific Ureteral Stents - Non-Tria
Number analyzed (Participants) | 215 | 144
Participants
  SADE Experienced | 2 | 3
  No SADEs Experienced | 213 | 141

3. Secondary Outcome: Quality of Life - Patient-Reported Outcomes
Description: Measurement System Patient Reported Outcomes Measurement Information System (PROMIS®) for subjects ≥18 years
  * Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Intensity 3a, score range for the change from Index procedure is -41.1 to 41.1
  * Patient-Reported Outcomes Measurement Information System (PROMIS) - Pain Interference 6b, score range for the change from Index procedure is -37.3 to 37.3
  Higher PROMIS score means worse quality of life
Time Frame: Change From Index Procedure to Stent Removal Visit; Change From Index Procedure to Post Stent Removal Visit Stent Removal: Typically, within 2 weeks to < 365 days from Index Procedure Post-Stent Removal: Typically, 3 - 12 weeks from Stent Removal
Population: Subjects who provided consent and for whom a Boston Scientific stent placement procedure was initiated were included.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Boston Scientific Ureteral Stents - Tria | Boston Scientific Ureteral Stents - Non-Tria
Number analyzed (Participants) | 215 | 144
score on a scale
  Pain Intensity Score Change From Index Procedure to Stent Removal Visit | -1.83 [-37.6 to 31.3] | 2.04 [-37.6 to 33.6]
  Pain Intensity Score Change From Index Procedure to Post Stent Removal Visit | -9.51 [-41.1 to 23.4] | -10.79 [-41.1 to 23.0]
  Pain Interference Score Change From Index Procedure to Stent Removal Visit | -2.76 [-37.2 to 37.2] | 2.25 [-34.0 to 34.0]
  Pain Interference Score Change From Index Procedure to Post Stent Removal Visit | -10.99 [-37.2 to 24.5] | -11.14 [-37.2 to 22.9]

4. Secondary Outcome: Stent Migration
Description: Stent Migration: Confirmed via imaging
Time Frame: 2 months to 15 Months
Population: Subjects who provided consent and for whom a Boston Scientific stent placement procedure was initiated were included. Number of units analyzed are for all stents implanted.
Measure: Count of Units; unit: Stent Implanted
Units Other Than Participants: Stent Implanted
Arm/Group | Boston Scientific Ureteral Stents - Tria | Boston Scientific Ureteral Stents - Non-Tria
Number analyzed (Participants) | 215 | 144
Number analyzed (Stent Implanted) | 263 | 165
Stent Implanted
  Stent Migration | 3 | 2
  No Stent Migration | 260 | 163

ADVERSE EVENTS:
Time Frame: up to 11 months. Adverse events were collected from the time of index procedure to end of the study for each subject enrolled.
Description: AE reporting includes; all- cause mortality, serious adverse events, and other adverse events (not including serious)
  SAE includes serious deterioration in health of subject, users or other persons; permanent impairment of a body structure or function including chronic diseases; fetal distress/death or physical or mental impairment.
Arm/Group | Boston Scientific Ureteral Stents - Tria | Boston Scientific Ureteral Stents - Non-Tria
All-Cause Mortality (participants affected / at risk) | 3/215 | 0/144
Serious Adverse Events (participants affected / at risk) | 9/215 | 5/144
Other Adverse Events (participants affected / at risk) | 57/215 | 40/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boston Scientific Ureteral Stents - Tria (N=215) | Boston Scientific Ureteral Stents - Non-Tria (N=144)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infections (Infections and infestations) | 0 (0) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Urinary Bladder Haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Valve Disease (Cardiac disorders) | 1 (1) | 0 (0)
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal Pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boston Scientific Ureteral Stents - Tria (N=215) | Boston Scientific Ureteral Stents - Non-Tria (N=144)
Flank Pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 16 (16)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bladder Spasm (Renal and urinary disorders) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1) | 4 (4)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition Disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition Urgency (Renal and urinary disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 15 (15) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Penile Pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Post Procedural Urine Leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 9 (9) | 13 (14)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Renal Colic (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal Pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Stent Placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urethral Pain (Renal and urinary disorders) | 6 (6) | 0 (0)
Urge Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT04197583/Prot_SAP_000.pdf